CLINICAL TRIAL: NCT03099967
Title: Cardiac Troponin T After Transcatheter Closure of the Interatrial Septum
Status: Completed | Type: Observational
Sponsor: Skane University Hospital (Other)
Responsible Party: Principal Investigator, Joanna Hlebowicz, MD, Associated Professor, Skane University Hospital
Other Study IDs: Interatrial septum 1
Record Dates: First submitted 2017-03-29; First posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Transcatheter closure of an atrial septal defect or patent foramen ovale. — In a prospective study in adults troponin T (TnT) serum concentrations were determined before and the day after transcatheter closure of an atrial septal defect (ASD) or patent foramen ovale (PFO).

SUMMARY:
To examine retrospectively whether transcatheter closure of the interatrial septum leads to myocardial injury and to determine the mechanism.

DETAILED DESCRIPTION:
In a prospective study in adults troponin T (TnT) serum concentrations were determined before and the day after transcatheter closure of an atrial septal defect (ASD) or patent foramen ovale (PFO).

ELIGIBILITY:
Inclusion Criteria:

* transcatheter ASD and PFO closure at the University Hospital of Lund, Sweden

Exclusion Criteria:

* missing TnT values

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fifty one patients who underwent transcatheter ASD and PFO closure (the University Hospital of Lund, Sweden) were studied retrospectively.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2005-01-01; Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
TnT changes | Blood samples for TnT were taken one day before intervention and one day after intervention.

IPD SHARING:
Plan to Share IPD: No